CLINICAL TRIAL: NCT03244657
Title: Phase IV Clinical Trial (STAR Study) Extension Study of Conbercept Ophthalmic Injection for Treatment of Polypoid Choroidal Vasculopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KH902-STE-CRP-1.2
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Polypoid Choroidal Vasculopathy (PCV)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Q12W group (Experimental)
  Interventions: Drug: conbercept ophthalmic injection （0.5mg）
- TAE group (Experimental)
  Interventions: Drug: conbercept ophthalmic injection （0.5mg）

INTERVENTIONS:
Drug: conbercept ophthalmic injection （0.5mg） — The target eye receives intravitreal injection of 0.5mg conbercept ophthalmic injection once every 12 weeks; if a subject meets "additional drug administration criteria" within 12 weeks between treatments, the subject can receive additional injection treatment
  Arms: Q12W group
Drug: conbercept ophthalmic injection （0.5mg） — In principle, the first administration time of the target eye uses the time determined by the assessment at end of STAR study; later, based on "treatment-extension drug administration criteria", an investigator determines next visit time/treatment interval according to assessment result at each visit.When a subject's visit/treatment interval extends to 12 weeks, an additional safety visit can be arranged if an investigator considers that there is suspicious active lesion; if assessment result at the safety visit meets "additional drug administration criteria", additional injection treatment can be given.
  Arms: TAE group

SUMMARY:
To explore efficacy and safety of 0.5 mg conbercept ophthalmic injection for long-term treatment of polypoid choroidal vasculopathy (PCV) subjects.

ELIGIBILITY:
Inclusion Criteria:

* (1) Sign the informed consent and be willing to receive follow-up at the time specified in the trial; (2) A subject who has completed all visits specified by STAR study protocol and who is within 3 months after end of the last visit (the following subjects can be included: during STAR study, an investigator decided to discontinue treatment from point of view of safety, but the risk factor has disappeared or become stable).

Note: Use the determined eye of STAR study as the target eye.

Exclusion Criteria:

* (1) A subject who actively withdrew from the study during STAR study; (2) The target eye or the body ever received other anti-VEGF drugs (such as Macugen, Lucentis, Avastin, Eylea, Zaltrap, etc.) from start of STAR study to before screening of this study.

  (3) In the target eye or the body, there is any following disease and condition: an investigator thinks that if the subject participates in this study, the disease and condition (such as: the target eye has history of vitrectomy; blood pressure control of a hypertension patient is not ideal [ after treatment of antihypertensive drugs, blood pressure is still ≥ 150/95 mmHg]; AIDS; malignant tumors; active hepatitis; renal failure; severe mental, neurological, cardiovascular, respiratory and other systemic diseases; ankylosing spondylitis; systemic lupus erythematosus; heart stent surgery; and the like) may cause the subject to be at relatively large risk; (4) A subject who ever had stroke, transient ischemic attack, myocardial infarction, or acute congestive heart failure and other cardiovascular events within 6 months before screening (5) A subject who participated in any drug (not including vitamins or minerals) clinical trial within 3 months (if the test drug has long half-life and 5 half-lives > 3 months, then 5 half-lives are taken) before screening;(6) Not take effective contraceptive measure; Note: The following conditions are not excluded. I. Amenorrhea for 12 months under natural condition; or, under natural condition, amenorrhea for 6 months, accompanied with follicle stimulating hormone level in serum > 40 mIU/ml; II. 6 weeks after bilateral oophorectomy with/without hysterectomy;

III. Use one or more of the following contraceptive methods:

* Sterilization (male with bilateral vasoligation, vasectomy)
* Hormone contraception (implantable type, patch type, oral administration type)
* Intrauterine device, double-barrier method IV. Be able to take reliable contraceptive measure throughout the study and insist on it till 30 days after discontinuation of the investigational drug (unacceptable contraceptive methods include: regular abstinence, i.e., depending on calendar, ovulatory period, body temperature measurement method and post-ovulation period method; coitus interruptus for extracorporeal spermiation). (7) Pregnant (in this trial, pregnancy is defined as positive urine pregnancy test), lactating females (8) A subject whom an investigator thinks needs to be excluded.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04-25 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
change of best corrected visual acuity (BCVA) | up to 40 week
  Assess mean of change of best corrected visual acuity (BCVA) compared with baseline in the target eyes (using the same target eyes as STAR study) of subjects at end of the extension study;
adverse events | up to 40 week
  Assess incidence and severity of adverse events in subjects.

SECONDARY OUTCOMES:
mean of change of BCVA | up to 40 week
  Assess mean of change of BCVA compared with that in STAR study baseline (before treatment) in the target eyes of subjects at end of the extension study
change of central retinal thickness (CRT) | up to 40 week
  Assess mean of change of central retinal thickness (CRT) compared with baseline in the target eyes of subjects at time of each visit till end of the extension study;
mean of change of lesion's maximum retinal thickness (MRT) | up to 40 week
  Assess mean of change of lesion's maximum retinal thickness (MRT), retinal pigment epithelium detachment's (PED) volume and thickness, polypoid lesion area, retinal hemorrhage area and other imaging indicators compared with baseline in the target eyes of subjects at end of the extension study;
average number of times of drug administration | up to 40 week
  Assess average number of times of drug administration in two groups of subjects during the extension treatment;

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Beijing Hospital, Beijin
  - The Chinese people's liberation army 474 hospital, Beijin
  - Beijing Tongren Hospital,Cmu, Beijing
  - Chinese Pla General Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People'S Hospital, Beijing
  - PEKING UNIVERSITY Third HOSPITAL, Beijing
  - Xiangya Hospital Central South University, Changsha
  - Hainan Eye Hospital of Zhongshan Ophthalmic Center, Sun Yat-sen University, Hainan
  - Hebei Eye Hospital, Hebei
  - The Second Hospital of Hebei Medical University, Hebei
  - Henan Province People's Hospital, Henan
  - The Second Hospital of Jilin University, Jilin
  - Lanzhou University Second Hospital, Lanzhou
  - Affiliated Eye Hospital of Nanchang University, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanjing
  - The First Affiliated Hospital With Nanjing Medical University, Nanjing
  - Eye&Ent Hospital of Fudan University, Shanghai
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Stu/Cuhk Joint Shantou International Eye Center, Shantou
  - Shanxi Eye Hospital, Shanxi
  - Shenzhen Eye Hospital, Shenzhen
  - Tianjin Medical University Eye Hospital, Tianjin
  - The Eye Hospital of Wmu Zhejiang Eye Hospital, Wenzhou
  - Renmin Hospital of Wuhan University, Wuhan
  - Xiamen Eye Centre of Xiamen University, Xiamen
  - Ningxia Peple'S Hospital, Yinchuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Zhejiang